CLINICAL TRIAL: NCT01612910
Title: A Pilot Study of BR-DIM in Women With Stage II-III, Triple Negative, and Androgen Receptor Positive, Invasive Breast Cancer, Who Have Residual Disease Following Surgical Resection After Neoadjuvant Chemotherapy
Brief Title: Oral Microencapsulated Diindolylmethane in Treating Patients With Stage II-III Triple Negative, Androgen Receptor Positive Breast Cancer Who Have Undergone Chemotherapy and Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Research cancelled.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Simon, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-111
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer Female
Keywords: estrogen receptor-negative breast cancer; HER2-negative breast cancer; progesterone receptor-negative breast cancer; recurrent breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; triple-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- microencapsulated diindolylmethane, lab. biomarker analysis (Experimental): Patients receive oral microencapsulated diindolylmethane orally (PO) twice a day (BID) for 1 year in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: oral microencapsulated diindolylmethane; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: oral microencapsulated diindolylmethane — Patients receive oral microencapsulated diindolylmethane orally (PO) twice a day (BID) for 1 year in the absence of disease progression or unacceptable toxicity
  Other Names: BioResponse DIM, BR-DIM
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This study is being done to find out whether a nutritional supplement, called BioResponse-DIM (BR-DIM [oral microencapsulated diindolylmethane]), improves the survival for women who have residual cancer cells following surgery after chemotherapy for breast cancer. BR-DIM is an active ingredient in cruciferous vegetables (broccoli, brussels sprouts and cauliflower). Consumption of these vegetables has been associated with a decreased risk in several cancers. Researchers also hope to find out whether different biomarkers (also called "markers") in the blood predict the chance of breast cancer returning. BR-DIM is thought to be effective in treating stage II-III breast cancer that is triple negative, AR positive (+), and where there is residual cancer cells in the breast after chemotherapy.

DETAILED DESCRIPTION:
Patients receive oral microencapsulated diindolylmethane orally (PO) twice daily (BID) for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a histologically or pathologically confirmed diagnosis of triple negative, AR positive invasive breast carcinoma (stage II or III) who have received neoadjuvant chemotherapy (anthracycline or taxane or both) who have residual disease in their breasts following surgical resection by lumpectomy or mastectomy; androgen receptor (AR) testing will be performed on all patients who have residual invasive breast cancer after neoadjuvant taxane and/or anthracycline for triple negative breast cancer; this will be done under institutional protocol approval; physicians of patients who have AR positive tumors will be notified by our research coordinator of the potential eligibility for this study
* Participants must have undergone definitive surgery with negative margins for breast cancer in the past 2 years and must have residual pathologic invasive disease in the primary breast or lymph nodes or both; at the time of protocol entry it will be determined under good medical practice that there is no evidence for metastatic disease; patients should have completed all radiation therapy if indicated at the time of study entry
* Patients must have a Zubrod performance status of 0-2
* Patients must consent to the serum and whole blood specimen submissions
* Patients must be able to take oral medications (patients with uncontrolled nausea, vomiting, diarrhea at baseline, lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, are excluded)

  * Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents; women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of this trial
  * Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
  * Granulocyte count > 1,500/mcL
  * Platelet count > 100,000/mcL
  * Bilirubin =< 3 x institutional upper limit of normal (IULN)
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5 x IULN
  * Serum creatinine =< 1.5 x IULN

Exclusion Criteria:

* Patients must not have a current active infection requiring systemic therapy
* Patients must not have had a cardiac event within 6 months prior to registration such as myocardial infarction (including severe/unstable angina), coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF), cerebrovascular accident or transient ischemic attack, or pulmonary embolism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS), defined as clear development of new sites of disease, measurable or non-measurable or death | From date of registration to date of first documentation of progression, up to 3 years
  Estimated using Kaplan-Meier methods with 95% confidence intervals.

SECONDARY OUTCOMES:
Association of serum BR-DIM levels and changes in correlative biomarkers with time to progression | Baseline
  Levels of correlative biomarkers explored using a proportional hazards model, with biomarkers parameterized as time-dependent covariates.
Association of serum BR-DIM levels and changes in correlative biomarkers with time to progression | Up to 3 years
  Levels of correlative biomarkers explored using a proportional hazards model, with biomarkers parameterized as time-dependent covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Simon, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute